CLINICAL TRIAL: NCT05860270
Title: The Effects of Oral Vitamin D Supplementation on the Prevention of Peritoneal Dialysis-related Peritonitis, a Multicenter Randomized Controlled Trial
Brief Title: Oral Vitamin D Supplementation Prevent Peritoneal Dialysis-related Peritonitis
Acronym: VD-PD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University Third Hospital (Other); Peking University People's Hospital (Other); Beijing Haidian Hospital (Other); Peking University Shenzhen Hospital (Other); Miyun District of Peking University First Hospital (Unknown); Beijing Fangshan District Hospital of Traditional Chinese Medicine (Unknown); Peking University International Hospital (Other); Beijing Tsinghua Changgeng Hospital (Other); Beijing Anzhen Hospital (Other); Capital Medical University (Other)
Responsible Party: Principal Investigator, Dong Jie, Director of PD center, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Vitamin D and Peritonitis
Record Dates: First submitted 2023-04-14; First posted 2023-05-16 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Peritoneal Dialysis-associated Peritonitis; Vitamin D Deficiency
Keywords: Peritoneal dialysis; Peritonitis; Cholecalciferol
MeSH Terms: conditions — Vitamin D Deficiency; Peritonitis | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Eligible patients on PD at one month after being cured from an episode of peritonitis will be enrolled and randomized 1:1 into two groups, includingthe intervention group administered Cholecalciferol (produced by Xymogen Company) 4000 U (2 capsules) per day, and the control group administered placebo 2 capsules per day.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Random number will be generated by statistician who is not involved in the study, and will be masked to all participants, caregivers, investigators and outcomes assessors. Only the drug dispensing personnel will have the decoding table. When an eligible patient is enrolled, he/she will be given a sequential patient number, according to block randomization. Such a patient number indicated its group allocation. The drug dispensing personnel will offer the corresponding drug, however with a random drug number. Serial Serum 25- hydroxy-Vitamin D levels, obtained every three months, will be declassified at the end of the study (24 months after enrollment), or till the occurrence of death, permanently transfer to hemodialysis, loss of follow-up, or withdrawal from the study, whichever comes first.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): Patients will be given Cholecalciferol (produced by Xymogen Company) 4000 U (2 capsules) per day
  Interventions: Drug: Cholecalciferol
- Control group (Placebo Comparator): Patients will receive placebo, 2 capsules per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — Patients in the intervention group will receive oral cholecalciferol 4000U per day.
  Other Names: Natural Vitamin D3
  Arms: Treatment group
Drug: Placebo — Patients in the control group will receive placebo 2 capsules per day.
  Arms: Control group

SUMMARY:
This is a multicenter randomized, placebo-controlled trial of Vitamin D supplementation in patients on peritoneal dialysis to determine whether oral administration of vitamin D3 after curing an episode of peritonitis could reduce the risk of subsequent peritoneal dialysis-related peritonitis.

DETAILED DESCRIPTION:
176 eligible patients on PD at one month after being cured from an episode of peritonitis will be enrolled and randomized into two groups, including the intervention group administered Cholecalciferol (produced by Xymogen Company) 4000 U (2 capsules) per day, and the control group administered placebo 2 capsules per day. All participants will be followed for 24 months, or till the occurrence of death, permanently transfer to hemodialysis, loss of follow-up, or withdrawal from the study, whichever comes first. The primary outcome is the occurrence of subsequent peritonitis. The study aims to identify whether oral administration of vitamin D3 after curing an episode of peritonitis could reduce the risk of subsequent peritoneal dialysis-related peritonitis.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable and receiving peritoneal dialysis for > 1 month
* Older than 18 years old
* Serum 25(OH)D < 30ng/ml
* Adequate dialysis on evaluation with weekly Kt/V ≥ 1.5, or (revised time: 2023-7-11) without clinical uremic symptoms

Exclusion Criteria:

* Receive Vitamin D2/D3 during the previous 1 month (revised time: 2023-7-11) ;
* History of allergic reaction to Cholecalciferol;
* Current or past malignant disease, active hepatitis or hepatic failure, active autoimmune disease, severe digestive malabsorption or an eating disorder, HIV/AIDS;
* Acute systemic infection, cardiovascular disease, surgery, or trauma in the last month;
* A high probability of receiving a kidney transplant or transferring to hemodialysis or drop-out due to socioeconomic causes within 6 months;
* History of kidney transplant;
* Hemodialysis combined with peritoneal dialysis currently;
* Pregnant or breastfeeding;
* Not suitable enrolled assessed by researchers, including patients who could not regular follow-up

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Hazard Ratio of Subsequent peritonitis | 24 months
  Risk of a subsequent episode of peritoneal dialysis related peritonitis in the interventional group compared with the control group measured by Hazard Ratio.

SECONDARY OUTCOMES:
rate of Systemic infection | 24 months
  Including respiratory infection, gastrointestinal infection, urinary system infection , skin infection etc.
rate of Technique failure due to peritonitis | 24 months
  Including peritonitis associated death (death within 30 days after peritonitis or death during hospitalization due to peritonitis), and transfer to hemodialysis due to uncured peritonitis.
rate of Death or transfer to hemodialysis with reasons other than peritonitis | 24 months
  Death or transfer to hemodialysis with reasons other than peritonitis

CONTACTS AND LOCATIONS:
Overall Officials: Jie Dong, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No